CLINICAL TRIAL: NCT03598660
Title: Role of Sorcin and Annexin A3 in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Breast cancer
Record Dates: First submitted 2018-07-08; First posted 2018-07-26 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer, SORCIN, Annexin A3
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast cancer patients: The present study will be carried on 50 breast cancer patients before surgery.
  The followings markers must be estimated:
  Sorcin gene expression using real time PCR and Annexin A3 serum mesurement using enzyme linked immuno sorbent assay (ELISA).
  Interventions: Genetic: Sorcin gene expression; Other: Annexin A3 serum mesurement
- Healthy controls: The present study will be carried on 15 age and sex matched controls.
  The followings markers must be estimated:
  Sorcin gene expression using real time PCR and Annexin A3 serum mesurement using ELISA.
  Interventions: Genetic: Sorcin gene expression; Other: Annexin A3 serum mesurement
- Benign breast diseases: The present study will be carried on 15 patients with benign breast diseases.
  The followings markers must be estimated:
  Sorcin gene expression using real time PCR and Annexin A3 serum mesurement using ELISA.
  Interventions: Genetic: Sorcin gene expression; Other: Annexin A3 serum mesurement

INTERVENTIONS:
Genetic: Sorcin gene expression — Sorcin gene expression Will be measured by real time PCR
Other: Annexin A3 serum mesurement — serum mesurement of Annexin A3 by enzyme linked immuno sorbent assay (ELISA)

SUMMARY:
Breast cancer (BC) is the most common female malignancy worldwide and the second leading cause of cancer death in women. One in eight women in the United States will develop the illness in their lifetimes. In Egypt, 37.7% of total cancer cases among women is breast cancer. A locally advanced disease is very common and total mastectomy is the most commonly performed surgery. Screening methods and adjuvant therapy following surgery led to a remarkable decrease in mortality.

Reliable prognostic and predictive markers are needed to guide the selection of the most appropriate adjuvant therapies for individual patients with breast cancer. In fact, a shift from defining the cancer patients who should receive chemotherapy on the basis of their prognostic characteristics to defining the patients who are likely to benefit most from this modality of adjuvant treatment is currently taking place. Understanding the molecular mechanisms underlying the spread of cancer cells to distant organs, therefore, is a prerequisite for the development of novel cancer therapies.

DETAILED DESCRIPTION:
Breast cancer is the most common female malignancy worldwide. Despite advances in cancer diagnosis and treatment in recent years, traditional treatments (radiotherapy, chemotherapy, and hormone therapy) are always limited by the resistance of some tumor cells, thus forcing researchers to continue to look for new therapeutic approaches and targets. Soluble resistance-related Calcium-binding protein (Sorcin) is a penta-EF hand calcium binding protein, which participates in the regulation of calcium homeostasis in cells and has molecular mass of 22 kDa. The EF-hand is a common helix-loop-helix structural motif used by proteins to bind calcium. Most proteins are endowed with an even number of EF-hands, which are usually structurally and functionally paired. The penta-EF hand (PEF) family includes sorcin, calpains, programmed cell death protein 6 (PDCD6), peflin and grancalcin.

High sorcin regulates the calcium channels and exchangers located at the plasma membrane and at the endo/sarcoplasmic reticulum (ER/SR) and allows high levels of calcium in the ER to be maintained, preventing ER stress and the unfolded protein response, and increases escape from apoptosis. The 18-kDa variant of sorcin is regulated by Tumor necrosis factor receptor-associated protein 1 (TRAP1), a mitochondrial anti-apoptotic protein upregulated in several human tumors which controls sorcin folding and expression. Conversely, sorcin silencing activates apoptotic proteases as caspase-3 and caspase-12 results in major defects in mitosis and cytokinesis, blocks cell cycle progression in mitosis, increases the number of rounded polynucleated cells and induces apoptosis and cell death shifting the equilibrium between cell life and cell death towards proliferation in MDR cancer cells overexpressing sorcin.

Sorcin is highly expressed in the heart, brain and breast and overexpressed in many cancer cells. The gene for sorcin (SRI) spans about 21.9 kb of human genomic DNA. The gene is located in chromosome 7q21. Sorcin gene is in the same amplicon as other genes involved in the resistance to chemotherapeutics in cancer cells (multi-drug resistance, MDR) such as the ATP-binding cassette (ABC) transporters ABCB4 and ABCB1 (Mdr1, or P-glycoprotein 1).

Annexins are a family of intracellular proteins that bind membrane phospholipids in a Calcium concentration-dependent manner. The human genome encodes for 12 different annexins varying in expression and distribution within the tissues. Some of these are ubiquitously expressed (A1, A2, A5, A6, and A7), while some are selective (A3, A8, A9, A10, and A13). Several annexins play important roles during tumor progression. However, little is known about the clinical implications and biological functions of Annexin A3 (ANXA3) in breast cancer. ANXA3 has a role in cell differentiation, cell migration, immune regulation.

The ANXA3 gene is located on human chromosome 4q13-q22 and encodes a protein of 323 amino acid residues. Annexin A3 participates in various tumor-associated biological processes, including tumor initiation, progression, metastasis and is associated with chemotherapy resistance.

ANXA3 is expressed and secreted by neoplastic mammary cells, and its inhibition halts migration in breast cancer cells. The expression of Annexin A3 in human breast carcinoma closely correlated with tumor size and axillary lymph node metastasis. Elevated serum levels of ANXA3 protein were due to its increased secretion from neoplastic breast cells into the systemic circulation. There is inverse correlation between Annexin A3 expression and overall breast cancer patient survival. Moreover, Annexin A3 might be a novel and potential prognostic marker for patients with breast cancer and is involved in regulating apoptosis by affecting the Bcl-2/Bax balance. It promote the transcription of the anti-apoptotic gene Bcl-2 and downregulate the proapoptotic gene BAX.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients before surgery who are admitted to the South Egypt Cancer Institute, Surgery Department, Assiut University

Exclusion Criteria:

* • Patients with malignancies elsewhere in the body.

  * Patients with chronic cardiac diseases.
  * Getting neoadjuvant chemotherapy.
  * Renal disease.
  * Neurodegenerative disease.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: breast cancer patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Role of SORCIN in patients with breast cancer | 1 year
  genetic expression of SORCIN new biomarker in breast cancer patients

SECONDARY OUTCOMES:
Role of annexin A3 biomarker in with breast cancer patients | 1 year
  serum measurement of annexin A3 in breast cancer patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeeneldin AA, Ramadan M, Elmashad N, Fakhr I, Diaa A, Mosaad E. Breast cancer laterality among Egyptian patients and its association with treatments and survival. J Egypt Natl Canc Inst. 2013 Dec;25(4):199-207. doi: 10.1016/j.jnci.2013.09.003. Epub 2013 Oct 25. PMID 24207092
- [Background] Cubasch H, Joffe M, Ruff P, Dietz D, Rosenbaum E, Murugan N, Chih MT, Ayeni O, Dickens C, Crew K, Jacobson JS, Neugut A. Breast conservation surgery versus total mastectomy among women with localized breast cancer in Soweto, South Africa. PLoS One. 2017 Aug 10;12(8):e0182125. doi: 10.1371/journal.pone.0182125. eCollection 2017. PMID 28797046
- [Background] Colotti G, Poser E, Fiorillo A, Genovese I, Chiarini V, Ilari A. Sorcin, a calcium binding protein involved in the multidrug resistance mechanisms in cancer cells. Molecules. 2014 Sep 5;19(9):13976-89. doi: 10.3390/molecules190913976. PMID 25197934
- [Background] Kim JY, Jung EJ, Park HJ, Lee JH, Song EJ, Kwag SJ, Park JH, Park T, Jeong SH, Jeong CY, Ju YT, Lee YJ, Hong SC. Tumor-Suppressing Effect of Silencing of Annexin A3 Expression in Breast Cancer. Clin Breast Cancer. 2018 Aug;18(4):e713-e719. doi: 10.1016/j.clbc.2017.11.009. Epub 2017 Nov 21. PMID 29217453